CLINICAL TRIAL: NCT04845256
Title: Evaluation of SOMAVAC 100 Sustained Vacuum System Versus Manual Suction Bulbs After Mastectomy With Immediate Breast Reconstruction
Brief Title: Evaluation of SOMAVAC 100 Sustained Vacuum System
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: PSG SOMAVAC
Record Dates: First submitted 2021-04-07; First posted 2021-04-14 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- SOMAVAC 100 Sustained Vacuum System: New sustained vacuum system
  Interventions: Device: SOMAVAC 100 Sustained Vacuum System

INTERVENTIONS:
Device: SOMAVAC 100 Sustained Vacuum System — Evaluate performance of sustained vacuum system compared to manual suction bulbs

SUMMARY:
The purpose of this research study is to compare the effectiveness of the Somavac 100 Sustained Vacuum System versus manual section bulbs after immediate breast reconstruction.

DETAILED DESCRIPTION:
Participants will undergo a screening that includes medical history review. Once screening is complete, participants will undergo immediate breast reconstruction per the surgeon's typical protocol. Surgeon will place up to two (2) drain(s) per breast as customary without changing their technique at the end of the surgical procedure. SOMAVAC® 100 Sustained Vacuum System will be attached to the end of the drain(s) on one side of the subject and standard of care manual suction bulbs attached to the other side. Subjects will return to the clinic every 72 hours for visits for the first 1 to 2 weeks, until the drain drops below 25mL, or as instructed by the physician. Each visit will take about 30 minutes. Subjects will have routine phone calls with the clinic to provide their drain output information to help determine when the drains should be removed. This is a study where the standard techniques of closed suction drainage are used for the removal of fluid from a surgical site. Hence, an increased risk related to post-operative care is not anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years or older; undergoing immediate pre-pectoral breast reconstruction after mastectomy (bilateral) with tissue expanders or implant
* Capable of providing informed consent
* Willingness to follow all study requirements including agreeing to attend all required follow-up visits and signs the informed consent.

Exclusion Criteria:

* Reconstruction is not post-mastectomy
* Pregnant or lactating females
* Patients needing more than 2 drains per breast
* Patients on steroids or other immune modulators known to impact healing
* Patients who are likely to not complete the study
* Patient who, in the opinion of the investigator, are unlikely to comply with the protocol
* Patients who have participated in this trial previously and who were withdrawn
* Patients with known allergies to contacting materials (i.e. latex, metal, etc.)
* Patients who received neoadjuvant chemotherapy or radiotherapy within the last 6 months
* Has any medical condition such as obesity (BMI>40), uncontrolled diabetes (HbA1c>7%) and/or immunosuppression.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Up to 25 patients (50 breasts) will be enrolled in this study who are undergoing immediate breast reconstruction after mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Impact of the SOMAVAC continuous suction device on postoperative fluid drainage after mastectomy reconstruction | Approximately 3 months
  Given that patients enrolled will have bilateral reconstruction, one side will have the SOMAVAC continuous suction device and the other side will have standard manual suction bulbs. The fluid drained on each side will be measured in milliliters over 24 hour periods, recorded, and analyzed for any difference.
The SOMAVAC continuous suction device and seroma development on reconstructed mastectomy patients | approximately 3 months
  Incidence of postoperative seromas requiring drainage will be recorded for each side. Fluid drained will be measured in milliliters and side differences will be analyzed for statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Brzezienski, MD, Principal Investigator — University of Tennessee College of Medicine Chattanooga, Department of Plastic Surgery
Locations (1):
- Plastic Surgery Group, Chattanooga, Tennessee, United States